CLINICAL TRIAL: NCT02692053
Title: Characterization of Hemostatic Disordres in Septic Shock: Searching for Biological Markers
Acronym: COASEPT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Diagnostica Stago (Industry)
Responsible Party: Principal Investigator, Pr Bruno LEVY, Professor, Central Hospital, Nancy, France
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-A00834-45
Record Dates: First submitted 2016-02-12; First posted 2016-02-25 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Blood Specimen Collection

ARMS (2):
- Patients with septic shock (Experimental)
  Interventions: Biological: blood sampling
- Blood samples from a historical cohort of healthy volunteers (Other)
  Interventions: Biological: blood sampling

INTERVENTIONS:
Biological: blood sampling — additional blood sampling (volume: 18 mL)

SUMMARY:
Sepsis induces hemostatic disorders due to the exessive or inappropriate activation of inflammation, which could lead either to hypercoagulability or hypocoagulability. It is currently not possible to determine the hemostatic status of a given patient. This instability of hemostatic system is not revealed by classical tests. Thus, a better characterization of hemostatic status could certainly improve patient care. This study aims at characterizing disorders of coagulation and fibrinolysis using "global" tests such as thrombin generation test or coagulolytic test. Furthermore, the association with biological markers of interest (such as microparticles, neutrophil elastase or histones) will be evaluated.

ELIGIBILITY:
Eligibility criteria for patients with septic schock

Inclusion Criteria:

* septic shock (Dellinger, 2013)
* age >18y
* hospitalized patients
* signature of an informed consent (emergency consent)
* affiliation to a social security regimen

Exclusion Criteria:

* pregnancy or breast-feeding women
* moribund patient
* oral anticoagulant therapy
* thrombophilia
* Minor patients
* Patients under tutelage

Eligibility criteria from subject without septic shock Subject blood samples without septic shock are collected from a historical healthy volunteers cohort.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Changes in endogenous thrombin potential as assessed by thrombin generation test | 48 hours
  thrombin generation will be measured using CAT method (fluorescence) in plasma from patients within 48 hours. Endogenous thrombin potential is defined as the area under the thrombin generation curve and will be compared with values obtained in healthy subjects

SECONDARY OUTCOMES:
Changes in Thrombin peak as assessed by thrombin generation test | 48 hours
  thrombin generation will be measured using CAT method (fluorescence) in plasma from patients within 48 hours. Thrombin peak is defined as the highest thrombin concentration derived from the thrombin generation curve and will be compared with values obtained in healthy subjects.
Changes in clot lysis time as assessed by clot lysis assay | 48 hours
  Clot lysis assay will, be performed in plasma from patients and will be compared with those obtained in healthy subjects.
Correlation of neutrophil elastase with changes in endogenous thrombin potential | 48 hours
  Neutrophil elastase will be measured in plasma from patients.
Correlation of cell-derived microparticles with changes in endogenous thrombin potential | 48 hours
  microparticles derived from leukocytes, erythrocytes, platelets and endothelial cells will be measured in plasma from patients by flow cytometry.
Correlation of circulating histones with changes in endogenous thrombin potential | 48 hours
  Circulating histones will be measured in plasma from patients